CLINICAL TRIAL: NCT05715619
Title: A Phase 1/2a Double-Blind, Randomized, Placebo-Controlled Trial to Assess the Safety and Efficacy of Oral Administration of the Phage Cocktail, VRELysin™, In Healthy And VRE-Colonized Subjects
Brief Title: Safety and Efficacy of Oral Administration of the Phage Cocktail, VRELysin™, In Healthy and VRE-Colonized Subjects
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intralytix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ITX/VL-001
Record Dates: First submitted 2023-01-06; First posted 2023-02-08 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Vancomycin-Resistant Enterococcal Colonization
Keywords: bacteriophage; phage; VRE; Enterococcus; vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Dose is 1mL of placebo given orally three times a day for 7 days (Phase 1) or 14 days (Phase 2a)
  Interventions: Other: Placebo
- VRELysin™ (Active Comparator): Dose is 1mL of bacteriophage preparation given orally three times a day for 7 days (Phase 1) or 14 days (Phase 2a)
  Interventions: Biological: VRELysin™

INTERVENTIONS:
Biological: VRELysin™ — A cocktail of lytic Enterococcus-specific bacteriophages orally administered with sodium bicarbonate solution
  Arms: VRELysin™
Other: Placebo — Placebo orally administered with sodium bicarbonate solution
  Other Names: Phosphate Buffered Saline
  Arms: Placebo

SUMMARY:
The study is a first-in-human Phase 1/2a randomized, double-blind, placebo-controlled trial to assess the clinical safety and efficacy of VRELysin in healthy and VRE-colonized adults.

DETAILED DESCRIPTION:
The purpose of this study is to determine if VRELysin is safe and effective in adults in a continuous Phase 1/2a trial. Phase 1 will asses the safety of VRELysin in healthy adults, while Phase 2a will evaluate the safety and efficacy of VRELysin in adults colonized with VRE in the gastrointestinal tract.

VRELysin is a collection of bacteriophages. Bacteriophages (or phages) are viruses that infect only bacteria. The phages in VRELysin infect a specific type of bacteria called Enterococcus, which can cause gastrointestinal infections. VRELysin is intended to significantly reduce or eliminate vancomycin-resistant Enterococcus (VRE) levels in the human gastrointestinal tract, which in turn, may prevent subsequent infection as well as nosocomial spread.

ELIGIBILITY:
PHASE 1 INCLUSION CRITERIA:

To be eligible to participate in the Phase 1 segment of the study, each subject must fulfill ALL of the following criteria:

1. Age 18 to 50 years old.
2. Body mass index (BMI) of ≥19 kg/m2 to ≤40 kg/m2.
3. Has the ability to understand the study procedures and risks involved with the study, voluntarily agrees to participate by giving written informed consent and is willing to adhere to dose and visit schedules. The subject must be able to read, understand, and complete questionnaires and memory aids.
4. Agrees not to enroll in another study of an investigational research agent during the study, with the exception of potentially lifesaving or coronavirus disease of 2019 (COVID-19)-related experimental treatments.
5. Good general health as shown by medical history, physical examination, and screening laboratory tests or clinical laboratory abnormalities per clinical judgment of Principal Investigator (PI).
6. Agrees not to donate blood or blood products during participation in the study or for 30 days after completion of study participation.
7. Has negative serology results for HIV, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
8. Female subjects must have a negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test at Screening and within 24 hours of initial treatment on Day 1.

   a. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records) are not required to undergo pregnancy testing.
9. Female subjects of reproductive potential must agree to use adequate contraception, defined as consistent and correct use of an FDA-recommended contraceptive method or combination of methods in accordance with the product label. For example:

   1. Barrier method (such as condoms, diaphragm, or cervical cap) used in conjunction with spermicide and another method, such as prescription hormonal contraceptive;
   2. Intrauterine device (IUD);
   3. Prescription hormonal contraceptive taken or administered via oral (pill), transdermal (patch) subdermal, or intramuscular route used in combination with another method, such as barrier methods;
   4. Total abstinence;
   5. Sterilization of a monogamous female participant's male partner prior to entry into the study.

   Note: periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
10. Female subjects must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required study visit is completed.
11. Male subjects must agree to use adequate contraception, defined as consistent and correct use of an FDA-recommended contraceptive method in accordance with the product label (see above), for the duration of the study and refrain from donating sperm during this period.

PHASE 1 EXCLUSION CRITERIA:

To be eligible to participate in Phase 1, subjects must NOT fulfill ANY of the following criteria:

1. Investigational research agents received within 30 days before first treatment.
2. Pregnant or breastfeeding.
3. Regular (no more than once a week) use of antidiarrheals, stool softeners, laxatives, antacids, or other agents to lower stomach acidity.
4. Use of oral or intravenous antimicrobials within 2 weeks of study start or planned use during active study phase. Topical treatments are allowed.
5. Proton pump inhibitors, H2 blockers or antacids within 48 hours prior to dosing or planned use during active study phase.
6. Abnormal bowel patterns, defined by <3 stools per week or >2 stools per day on average over the past 6 months.
7. History of diarrhea in the 7 days prior to treatment. Outpatient diarrhea is defined as ≥ 3 unformed (Grade 3 or greater) loose stools in 24 hours.
8. Use of oral supplemental probiotics in the form of pills or tablets within 2 weeks of study start or planned use during active study phase.
9. History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up).
10. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes, but is not limited to:

    1. Any contraindication to repeated blood draws;
    2. A condition or process for which signs or symptoms could be confused with reactions to treatment;
    3. Any of the following in the past 10 years: Crohn's disease, ulcerative colitis, irritable bowel disease, celiac disease, stomach, or intestinal ulcers, or 2 or more episodes of inflammatory arthritis (joint pain and swelling);
    4. Bacterial infection at time of enrollment;
    5. Blood in stool on >2 occasions (other than small amounts from straining) in past 12 months;
    6. Recurrent diarrhea (>5 episodes in past 6 months, each lasting >3 days or more).
11. History of excessive alcohol consumption or drug dependence within last 3 years.
12. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety, or a subject's ability to give informed consent.
13. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
14. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
15. Malignancy (Not excluded from participation: subject who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study).
16. Seizure disorder/epilepsy: History of seizure(s) within past 3 years. Also exclude if subject has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
17. Asplenia: any condition resulting in the absence of a functional spleen.
18. History of chronic gastrointestinal illness, including severe dyspepsia, lactose intolerance, or other significant gastrointestinal tract disease (e.g., irritable bowel syndrome/disease, inflammatory bowel syndrome, gastric ulcer disease, Crohn's disease).
19. Any other criteria which, in the Investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study, or the results of the study.
20. Known allergy or hypersensitivity to an excipient in the study drug or placebo.

PHASE 2A INCLUSION CRITERIA:

To be eligible to participate in the Phase 2a segment of the study, each subject must fulfill ALL of the following criteria:

1. Age 18 to 50 years old.
2. BMI of ≥19 kg/m2 to ≤40 kg/m2.
3. Has the ability to understand the study procedures and risks involved with the study, voluntarily agrees to participate by giving written informed consent and is willing to adhere to dose and visit schedules. The subject must be able to read, understand, and complete questionnaires and memory aids.
4. Agrees not to enroll in another study of an investigational research agent during the study, with the exception of potentially lifesaving or COVID-19-related experimental treatments.
5. Agrees not to donate blood or blood products during participation in the study or for 30 days after completion of study participation.
6. Has negative serology results for HIV, HBsAg, and HCV antibody.
7. Has 2 consecutive positive VRE stool cultures (at least 7 days apart) that are susceptible to VRELysin. The second stool culture must be within 7 days of randomization.
8. Able to tolerate and take oral medication at time of randomization.
9. Female subjects must have a negative serum or urine β-HCG pregnancy test at Screening and within 24 hours of initial treatment on Day 1.
10. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records) are not required to undergo pregnancy testing.

    1. Female subjects of reproductive potential must agree to use adequate contraception, defined as consistent and correct use of an FDA-recommended contraceptive method or combination of methods in accordance with the product label. For example:
    2. Barrier method (such as condoms, diaphragm, or cervical cap) used in conjunction with spermicide and another method, such as prescription hormonal contraceptive;
    3. IUD;
    4. Prescription hormonal contraceptive taken or administered via oral (pill), transdermal (patch) subdermal, or intramuscular route used in combination with another method, such as barrier methods;
    5. Total abstinence;
    6. Sterilization of a monogamous female participant's male partner prior to entry into the study.

    Note: periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
11. Female subjects must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required study visit is completed.
12. Male subjects must agree to use adequate contraception, defined as consistent and correct use of an FDA-recommended contraceptive method in accordance with the product label (see above), for the duration of the study and refrain from donating sperm during this period.

PHASE 2A EXCLUSION CRITERIA:

To be eligible to participate in Phase 2a, subjects must NOT fulfill ANY of the following criteria:

1. Investigational research agents received within 30 days before first treatment.
2. Pregnant or breastfeeding.
3. Regular (no more than once a week) use of antidiarrheals, stool softeners, laxatives, antacids, or other agents to lower stomach acidity.
4. Use of oral or intravenous antimicrobials within 2 weeks of study start or planned use during active study phase. Topical treatments are allowed.
5. Proton pump inhibitors, H2 blockers or antacids within 48 hours prior to dosing or planned use during active study phase.
6. Abnormal bowel patterns, defined by <3 stools per week or >2 stools per day on average over the past 6 months.
7. History of diarrhea in the 7 days prior to treatment. Outpatient diarrhea is defined as ≥3 unformed (Grade 3 or greater) loose stools in 24 hours.
8. Taking supplemental probiotics in the form of pills or tablets within 2 weeks.
9. History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up).
10. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    1. Any contraindication to repeated blood draws;
    2. A condition or process for which signs or symptoms could be confused with reactions to treatment;
    3. Any of the following in the past 10 years: Crohn's disease, ulcerative colitis, irritable bowel disease, celiac disease, stomach, or intestinal ulcers;
    4. Blood in stool on >2 occasions (other than small amounts from straining) in past 12 months;
    5. Recurrent diarrhea (>5 episodes in past 6 months, each lasting >3 days or more);
    6. Requires hemodialysis.
11. History of excessive alcohol consumption or drug dependence within last 3 years.
12. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety, or a subject's ability to give informed consent.
13. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
14. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
15. Malignancy (Not excluded from participation: subject who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study).
16. Seizure disorder/epilepsy: History of seizure(s) within past 3 years. Also exclude if subject has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
17. Asplenia: any condition resulting in the absence of a functional spleen.
18. History of chronic gastrointestinal illness, including severe dyspepsia, lactose intolerance, or other significant gastrointestinal tract disease (e.g., irritable bowel syndrome, inflammatory bowel syndrome, gastric ulcer disease).
19. Known allergy or hypersensitivity to an excipient in the study drug or placebo.
20. Patients with active infection, a systemic infection requiring treatment, or any other unstable medical condition that could interfere with the study objectives.
21. Any other criteria which, in the Investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study, or the results of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number and Severity of Solicited and Unsolicited Adverse Reactions | Up to 36 days
  Number of subjects reporting solicited and unsolicited AEs, laboratory measures of safety, and AEs (up to Day 22) and serious adverse events (SAEs) (up to day 36) following treatment with VRELysin or placebo
Phase 2a: Number and Severity of Solicited and Unsolicited Adverse Reactions | Up to 180 days
  Number of subjects reporting solicited and unsolicited AEs, laboratory measures of safety and AEs (up to Day 29) and SAEs (up to Day 180) following treatment with VRELysin or placebo

SECONDARY OUTCOMES:
Phase 2a: Change in Number of VRE Organisms Secreted in Stool | up to Day 15
  Change from baseline to Day 15 in log10-transformed colony forming units (CFUs) of VRE shedding in stool samples following treatment with VRELysin or placebo
Phase 2a: Number of VRE Organisms Secreted in Stool at Day 15 | Day 15
  Quantitative (log10-transformed CFUs) assessment of VRE shedding in stool samples following treatment with VRELysin or placebo
Phase 2a: Decolonization of VRE in Stool at Day 15 | Day 15
  Day 15 decolonization defined as CFUs below the lower limit of quantitation
Phase 2a: Number of VRE Organisms Secreted in Stool at Day 29 | Day 29
  Quantitative (log10-transformed CFUs) assessment of VRE shedding in stool samples following treatment with VRELysin or placebo
Phase 2a: Number of VRE Organisms Secreted in Stool at Day 90 | Day 90
  Quantitative (log10-transformed CFUs) assessment of VRE shedding in stool samples following treatment with VRELysin or placebo

OTHER OUTCOMES:
Phase 1: Number of VRE-specific Bacteriophage Shed in Blood and Stool | up to Day 8
  Quantitation (mean, median and geometric mean plaque forming units [PFUs]) of bacteriophage shedding in blood and stool samples following treatment with VRELysin or placebo using plaque forming assays
Phase 1: Effect on Gut Microbiome Community States | up to Day 8
  Assess the effect of oral phage administration on the gut microbiome (e.g., mean species diversity) in stool samples following administration of VRELysin or placebo using next generation sequencing
Phase 2a: Number of VRE-specific Bacteriophage Shed in Blood and Stool | up to Day 29
  Quantitation (mean, median and geometric mean PFUs) of bacteriophage shedding in blood and stool samples following treatment with VRELysin or placebo using plaque forming assays
Phase 2a: Effect on Gut Microbiome Community States | up to Day 90
  Assess the effect of oral phage administration on the gut microbiome (e.g., mean species diversity) in stool samples following administration of VRELysin or placebo using next generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Minh-Hong Nguyen, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No